CLINICAL TRIAL: NCT04907903
Title: RinasciMENTE, An Internet-Based Self-Help Intervention for People With Psychological Distress Due to Coronavirus-19: Study Protocol of a Randomized Controlled Trial
Brief Title: RinasciMENTE, An Internet-Based Self-Help Intervention for People With Psychological Distress Due to COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Bar-Ilan University, Israel (Other); Istituto Auxologico Italiano (Other); Linkoeping University (Other Government); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Vanessa Bertuzzi, PhD Student, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-21
Record Dates: First submitted 2021-04-07; First posted 2021-06-01 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Psychological Disease
Keywords: COVID-19; internet-based intervention; cognitive-behavioral therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RinasciMENTE (Experimental): Participants will receive the internet-based intervention.
  Interventions: Other: internet-based intervention
- Waiting-list (No Intervention): Participants will no receive the internet-based intervention.

INTERVENTIONS:
Other: internet-based intervention — Intervention consists in 8 weekly online cognitive-behavioral modules (for a total duration of 2 months).
  Arms: RinasciMENTE

SUMMARY:
This study aims is the evaluation of the efficacy and feasibility of RinasciMENTE, the Randomized Controlled Clinical Trial compared with a waiting list control group.

DETAILED DESCRIPTION:
A sample of 128 participants, who experience psychological discomfort due to COVID-19, will be recruited. After initial screening, participants will be randomly assigned to either an experimental group or a waiting list group. Measures will be taken at the baseline (T0), at the end of the treatment (T1) and 12 months follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over and both gender
* Italian mother-tongue
* Score 14 or less on Patients Health Questionnaire-9 (PHQ-9)
* Internet access and basic informatic ability to navigate the internet platform
* Must be able to complete a phone interview

Exclusion Criteria:

* Having severe and mental impairments, psychiatric condition and neurological disorder
* Not be able to use a computer or do not have internet access
* Not be able to complete a phone interview
* Score 15 or more on PHQ-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Outcome Questionnaire (OQ-45) | Baseline, 2 months follow-up, 12 months follow-up
  It measures the changes in adult patients thanks to intervention.

SECONDARY OUTCOMES:
Perceived stress scale (PSS) | Baseline, 2 months follow-up, 12 months follow-up
  It evaluates the perceived stress by person
Emotional regulation questionnaire (ERQ) | Baseline, 2 months follow-up, 12 months follow-up
  It measures how respondents regulate their emotions through two dimensions: cognitive revaluation and expressive suppression.
Depression Anxiety Stress Scales-Short Version (DASS-21) | Baseline, 2 months follow-up, 12 months follow-up
  It allows to observe three dimensions (depression, anxiety and stress)
Fear of COVID-19 Scale (FCV-19S) | Baseline, 2 months follow-up, 12 months follow-up
  It evaluates how subjects show fear relative to the recent pandemic of Coronavirus
General Self-efficacy Scale (GSES) | Baseline, 2 months follow-up, 12 months follow-up
  It evaluates the confidence of subjects in their ability to cope with a variety of difficult or stressing situations.
World Health Organization Quality of Life (WHOQOL)-BREF | Baseline, 2 months follow-up, 12 months follow-up
  It detects four dimensions of quality of life: physical health, psychological health, social relations and environment.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04907903/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04907903/ICF_001.pdf